CLINICAL TRIAL: NCT01236118
Title: An Open-Label Extension Study to Evaluate Safety and Tolerability of Multiple Subcutaneous Doses of LY2439821 in Japanese Patients With Rheumatoid Arthritis on Concomitant Methotrexate
Brief Title: A Study of LY2439821 in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13625; I1F-JE-RHAM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 30 milligrams (mg) LY2439821 (Experimental): Participants will start receiving LY2439821 30 mg once every week for the first 3 doses and then once every 2 weeks until week 44. Investigators or its designees will increase the LY2439821 dose to 160 mg at any visit once the safety of LY2439821 180 mg is confirmed by the Data Review Meeting in Study I1F-JE-RHAL (NCT01253265).
  Interventions: Drug: LY2439821
- 80 mg LY2439821 (Experimental): Participants will start receiving LY2439821 80 mg once every week for the first 3 doses and then once every 2 weeks until week 44. Investigators or its designees will increase the LY2439821 dose to 160 mg at any visit once the safety of LY2439821 180 mg is confirmed by the Data Review Meeting in Study I1F-JE-RHAL (NCT01253265).
  Interventions: Drug: LY2439821
- 160 mg LY2439821 (Experimental): Participants will start receiving LY2439821 160 mg once every 2 weeks for the first 3 doses and then once every 4 weeks until Week 44.
  Interventions: Drug: LY2439821

INTERVENTIONS:
Drug: LY2439821 — Administered subcutaneously

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of LY2439821 subcutaneously administered for 48 weeks in Japanese participants with rheumatoid arthritis who have completed Study I1F-JE-RHAL (NCT01253265).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have received 7 injections of LY2439821 subcutaneously in the 30-, 80-, or 180-mg dose cohorts, or 11 injections in the 240-mg loading dose/120-mg once-a-week maintenance dose group, and completed the follow-up period (14 weeks) in Study I1F-JE-RHAL ((NCT01253265).
* Ambulatory male or female participants.

  * Male participants: Agree to use a reliable method of birth control during the study including barrier contraceptives or a monogamous relationship with a partner who is not child bearing.
  * Female participants: Are women who test negative for pregnancy at the time of entry based on a pregnancy test and are not breast feeding. Women of child bearing potential must agree to use a reliable method of birth control during the study.
* Participants who have been treated with methotrexate (MTX) throughout Study I1F-JE-RHAL (NCT01253265). Bucillamine, sulfasalazine and/or hydroxychloroquine are allowed to be administered in addition to MTX. In such a case, the participant needs to have been on a stable dose of the drug(s) throughout Study I1F-JE-RHAL (NCT01253265) and I1F-JE-RHAM.
* Participants who have given written informed consent approved by the Sponsor and the Institutional Review Board (IRB) governing the investigational site.

Exclusion Criteria:

* Participants who have had, during Study I1F-JE-RHAL (NCT01253265), any safety event including having a recent, ongoing, or serious infection, a serious drug reaction, or any adverse event (AE) that caused discontinuation from treatment , that in the opinion of the investigator poses an unacceptable risk to participation in this study.
* Participants who have any of the following abnormalities of clinical laboratory test results by Week 26 of Study I1F-JE-RHAL (NCT01253265):

  * Absolute neutrophil count <1000 cells/microliters (μL);
  * Lymphocyte count <500 cells/μL; or
  * White Blood Cells (WBC) count <2000 cells/μL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants must have completed Study I1F-JE-RHAL (NCT01253265) to meet the enrollment criteria of this study.
Groups:
- 30 mg LY2439821: Included participants from 30 milligrams (mg) group of Study I1F-JE-RHAL (NCT01253265). Participants received 30 mg LY2439821 subcutaneous injection once every week (Q1W) for the first 3 doses and once every 2 weeks (Q2W) until the safety data was confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection once every 4 weeks (Q4W) until Week 44.
- 80 mg LY2439821: Included participants from 80 mg group of Study I1F-JE-RHAL (NCT01253265). Participants received 80 mg LY2439821 subcutaneous injection Q1W for the first 3 doses and Q2W until the safety data was confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection Q4W until Week 44.
- 160 mg LY2439821: Included participants from either 30 mg or 80 mg group and started after the safety of 180 mg dose was confirmed in the Study I1F-JE-RHAL (NCT01253265). Participants received 160 mg LY2439821 subcutaneous injection Q2W for the first 3 doses then Q4W until Week 44.
Period: Overall Study
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 160 mg LY2439821
Started | 6 | 5 | 17
Completed | 4 | 4 | 14
Not Completed | 2 | 1 | 3
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 30 mg LY2439821: Included participants from 30 mg group of Study I1F-JE-RHAL (NCT01253265). Participants received 30 mg LY2439821 subcutaneous injection Q1W for the first 3 doses Q2W until the safety data was confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection Q4W until Week 44.
- 80 mg LY2439821: Included participants from 80 mg group of Study I1F-JE-RHAL (NCT01253265). Participants received 80 mg LY2439821 Q1W subcutaneous injection for the first 3 doses and then Q2W until the safety data was confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection Q4W until Week 44.
- 160 mg LY2439821: Included participants from either 30 mg or 80 mg group and started after the safety of 180 mg dose was confirmed in the Study I1F-JE-RHAL (NCT01253265). Participants received 160 mg LY2439821 Q2W subcutaneous injection for the first 3 doses then Q4W until Week 44.
- Total: Total of all reporting groups
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 160 mg LY2439821 | Total
Number analyzed (Participants) | 6 | 5 | 17 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (15.0) | 61.2 (8.1) | 57.6 (11.4) | 57.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 10 | 18
  Male | 3 | 0 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 17 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 5 | 17 | 28
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 5 | 17 | 28
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 54.23 (9.69) | 54.12 (7.66) | 61.25 (15.55) | 58.47 (13.48)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 161.62 (9.62) | 152.34 (6.20) | 159.52 (8.87) | 158.69 (8.90)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — BMI is an estimate of body fat based on body weight in kilograms divided by height squared in meters.
  kilograms per square meter (kg/m^2) | 20.68 (2.37) | 23.38 (3.50) | 23.95 (5.28) | 23.15 (4.60)
Weekly Dose of Methotrexate (MTX) [Mean (Standard Deviation); unit: milligrams per week (mg/week)] | 9.08 (1.86) | 8.40 (0.89) | 8.35 (0.79) | 8.52 (1.10)
Number of Participants Given Doses in Study I1F-JE-RHAL (NCT01253265) [Number; unit: participants]
  LY2439821 | 4 | 4 | 14 | 22
  Placebo | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) [Clinically Significant Events]
Description: Data presented are the number of participants who experienced 1 or more AEs (all causalities and drug-related) and serious AEs (SAEs). A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this report.
Time Frame: Baseline through study completion (up to Week 56)
Population: All enrolled participants.
Measure: Number; unit: participants
Groups:
- 30 mg LY2439821: Included participants from 30 mg group of Study I1F-JE-RHAL (NCT01253265). Participants received 30 mg LY2439821 subcutaneous injection Q1W for the first 3 doses and Q2W until the safety data confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection Q4W until Week 44.
- 80 mg LY2439821: Included participants from 80 mg group of Study I1F-JE-RHAL (NCT01253265). Participants received 80 mg LY2439821 Q1W subcutaneous injection for the first 3 doses and Q2W until the safety data was confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection Q4W until Week 44.
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 160 mg LY2439821
Number analyzed (Participants) | 6 | 5 | 17
participants
  AEs (All Causalities) | 6 | 5 | 16
  AEs (Drug-Related) | 3 | 4 | 7
  SAEs | 1 | 0 | 2

ADVERSE EVENTS:
Groups:
- 30 mg LY2439821: Included participants from 30 mg group of Study I1F-JE-RHAL (NCT01253265). Participants received 30 mg LY2439821 subcutaneous injection Q1W for the first 3 doses and Q2W until the safety data was confirmed to increase the dose. Dose was increased to 160 mg once safety of 180 mg dose was confirmed in Study I1F-JE-RHAL (NCT01253265). Participants then received 160 mg LY2439821 subcutaneous injection Q4W until Week 44.
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 160 mg LY2439821
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5 | 2/17
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg LY2439821 (N=6) | 80 mg LY2439821 (N=5) | 160 mg LY2439821 (N=17)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg LY2439821 (N=6) | 80 mg LY2439821 (N=5) | 160 mg LY2439821 (N=17)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Administration site reaction (General disorders) | 0 (0) | 0 (0) | 1 (13)
Injection site erythema (General disorders) | 1 (17) | 1 (11) | 1 (2)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Systemic mycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Hepatitis b dna assay positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Skin operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days